CLINICAL TRIAL: NCT03209557
Title: Pilot Trial Testing Feasibility and Effectiveness of Using SmokeBeat to Monitor and Increase Smoking Abstinence in Pregnant Women
Brief Title: Pilot Trial of Using SmokeBeat to Monitor and Increase Smoking Abstinence in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Alison Buttenheim, Assistant Professor of Nursing, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 827096
Record Dates: First submitted 2017-06-14; First posted 2017-07-06 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Tobacco Use Cessation; Pregnancy Related
Keywords: Mobile Technology; Sociobehavioral
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): 25 pregnant women will be enrolled and provided with usual care through Healthy Beginnings or NFP but will not receive a smartwatch or the active intervention. Smoking behavior will be measured by self-report and sample testing for the duration of the trial. Self-reported smoking status will be collected weekly. Sample testing will occur weekly and will be identical to the intervention group. They will be compensated for sample collection and survey completion.
- SmokeBeat Intervention (Experimental): 25 pregnant women will be enrolled and provided with a smartwatch. The smartwatch SmokeBeat application will be active. Smoking behavior will be measured by the smartwatch for the duration of the trial. Self-reported smoking status will be collected weekly. Sample testing will occur weekly.
  A second phase of the trial was initiated to evaluate a new watch. The smoking habits of participants who are receiving financial incentives to wear the watch are being compared to participants who are being given financial incentives for every day they go without smoking.
  A third phase of the trial was initiated to evaluate efficacy of larger financial incentives. All participants are incentivized to wear the watch, with the experimental arm also incentivized to abstain from smoking.
  Interventions: Other: SmartWatch SmokeBeat Application

INTERVENTIONS:
Other: SmartWatch SmokeBeat Application — The SmokeBeat app is a digital health app that allows for the user to monitor their smoking behavior in real time, set smoking cessation goals, and allows investigators, doctors and others using the app with participants to send messages directly related to smoking behavior. The SmokeBeat app, developed by Somatix Inc., will collects time-stamped on hand movements associated with smoking behavior. Participants will receive notifications on their phone and smartwatch when a smoking bout has been detected. In addition this app will deliver daily text messages aimed at improving quit rates among participants. We will be able to create the types of messaging we want to send and to modify when these messages will be sent to all participants. http://somatixinc.com/smokebeat/
  Arms: SmokeBeat Intervention

SUMMARY:
Investigators will assess the feasibility of implementing a randomized control trial of a behavioral intervention that uses smartwatch technology to monitor smoking behavior with texts aimed at reducing smoking in pregnant women who smoke. Investigators will compare the cessation rate of pregnant women who receive usual care through programs aimed at reducing smoking with pregnant women who receive usual care and are using the SmokeBeat app with a smartwatch.

DETAILED DESCRIPTION:
Somatix, LGH, and the Center for Health Incentives and Behavioral Economics of the University of Pennsylvania (CHIBE) will collaborate in using the unique smoking recognition technology of SmokeBeat app to track and analyze the smoking habits of LGH target smoking population. The target population for the SmokeBeat pilot is low-income pregnant women who smoke. This will enable us to gain insights on this target population and reach higher effectiveness of smoking cessation. Each participant will be enrolled in the trial for 12 weeks. Women randomized to the intervention arm will be given an Asus Zenwatch 2 smartwatch and a smartphone data plan for the duration of the study. Women assigned to the control group will be given the same smartwatch to keep following their participation in the trial. The tentative start date is June 2017.

After completing the consent participants will be randomized to one of two study arms. The control arm will consist of 25 pregnant women. Each will be provided with usual care through Healthy Beginnings or NFP but will not receive a smartwatch or the active intervention. Smoking behavior will be measured by self-report and sample testing for the duration of the trial. Self-reported smoking status will be collected weekly. Sample testing will occur weekly and will be identical to the intervention group. Following their completion of this trial they will receive a smartwatch as well. The intervention arm will consist of 25 pregnant women. Each will be enrolled and provided with a smartwatch. The SmokeBeat app will be active. Smoking behavior will be measured by the smartwatch for the duration of the trial. Self-reported smoking status will be collected weekly. Sample testing will occur weekly. All participants assigned to the intervention arm will be allowed to keep the smartwatch for their participation and be provided with a smartphone data plan for the duration of the study.

Two types of tests will be conducted with each participant, regardless of self-reported quit status. NicAlert strip tests (semi quantitative test) will be used to test saliva cotinine during weeks 2, 3, 5, 6, 8, 9, 11, and 12 of the participant's participation. This test will provide us with an accurate indicator of whether or not women have quit smoking while reducing the cost of the pilot study. A quantitative liquid chromatography cotinine test conducted by ARUP Labs will be used to test urine during weeks 1, 4, 7, and 10 for all women regardless of self-reported and smartwatch smoking status. This test, while more expensive, will provide us with the concentration of cotinine for each participant. This number can be directly compared to the self-reported and smartwatch reported number of cigarettes smoked as a way to validate self-report and smartwatch accuracy even when a participant has not quit smoking completely.

The main research instruments will consist of questionnaires on a subjects smoking habits and psychological tests that will help evaluate which types of patients are most able to quit smoking. All participants will be asked to complete an intake questionnaire at baseline (estimated length 15 minutes) and an exit questionnaire at the end of study participation 3 months after they start in the program (estimated length 15 minutes). Investigators will examine whether baseline values and/or changes during 3 months in these variables confound, causally mediate, or modify the effects of the intervention on quit rates. (a) Standard questionnaires will be administered to collect the following information: demographics (age, gender, ethnicity, marital status, and education), number of years of smoking, number of prior quit attempts, duration of previous abstinence periods, and current smoking rate. Nicotine dependence will be measured by the modified Fagerström Test for Nicotine Dependence (FTND), a 6-item measure of nicotine dependence. The FTND has satisfactory internal consistency (Cronbachs alpha=0.64) and high test-retest reliability (r=0.88).3 Heavy smokers are at highest risk for smoking related illnesses. Some but not all studies suggest that heavier smokers have lower quit rates. Investigators will evaluate whether FTND score either confounds or modifies the effects of the intervention. (b) Investigators will measure smoker's baseline readiness to quit using the Prochaska Stage of Change. (c) Investigators will assess participant's types and locations of jobs and whether they are exposed to smoking at home or in the workplace. (d) Participants use, durations, and doses of nicotine replacement therapy, varenicline, and buproprion will be assessed throughout the study. Participants will be asked to not use Nicotine patches or gum during the course of the study so that it will not interfere with weekly testing for smoking abstinence. (e) Time (or delay) discounting. Time discounting (known interchangeably as present-biased preferences or delay discounting) is a measure of impulsivity that reflects people's tendencies to discount the value of a reward as a function of how far in the future it would be received. People who smoke and use other drugs have steeper delayed discounting functions, meaning they have stronger present biased preferences. This is expected because smoking, like other unhealthy behaviors, entails immediate gratifications in exchange for future health problems. This also suggests that provision of early rewards, such as payments, might more effectively promote smoking cessation than interventions focusing on future rewards such as long-term health benefits, and that this effect might be strongest among those with the steepest discounting functions. Consistent with prior work, investigators will use a 7-item monetary choice questionnaire that defines ranges of delayed discounting by fitting a hyperbolic function to participants expressed preferences for smaller immediate versus larger delayed rewards. Information will also be collected weekly from participants on withdrawal and craving for nicotine as well as self-reported number of cigarettes per week. Investigators will also administer a 5 question weekly survey that addresses weekly levels of cravings, stress, social support, and asks about current cigarette use. All questions will be rated on a Likert scale, except for the number of cigarettes smoked, that will be an estimate of use.

The SmokeBeat app is a digital health app that allows for the user to monitor their smoking behavior in real time, set smoking cessation goals, and allows investigators, doctors and others using the app with participants to send messages directly related to smoking behavior. The SmokeBeat app, developed by Somatix Inc., will collects time-stamped on hand movements associated with smoking behavior. Participants will receive notifications on their phone and smartwatch when a smoking bout has been detected. In addition this app will deliver daily text messages aimed at improving quit rates among participants. Investigators will be able to create the types of messaging they want to send and to modify when these messages will be sent to all participants. http://somatixinc.com/smokebeat/.

A second pilot were begun in the summer of 2018. Intervention participants were offered a monetary reward for each day they went without smoking. Control participants were offered a financial incentive to wear the watch. In the fall of 2018 a third will start with an increase in the financial incentive, and a new smart band model.

A third pilot was started in the winter of 2018/2019. New participants were recruited, who were then randomized to one of two arms. Both arms were given smartbands that tracked their smoking use. Participants in the control arm were offered financial incentives for every day that they consistently wore the smartband. Participants in the experimental arm were offered financial incentives for consistently wearing the smartband and abstaining from smoking. All participants completed remote nicotine testing and survey questionnaires with study personnel via video chat. Five weekly video chats are scheduled with participants.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or within 3 weeks postpartum
* Self-reported smoking
* Part of the Nurse Family Partnership or Healthy Beginnings
* Uses an Android smart phone

Exclusion Criteria:

* Does not speak English
* Not interested in wearing a smart watch for 12 weeks

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Based on whether someone is currently pregnant or within 3 weeks post-partum
Enrollment: 32 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Smoking cessation rate biochemical verification | 12 weeks
  Quit rates in control vs. intervention group as determined by weekly cotinine testing.
Smoking cessation rate smartwatch | 12 weeks
  Quit rates in control vs. intervention group as measured by the smartwatch.

SECONDARY OUTCOMES:
Desire to quit | 12 weeks
  We will compare the self-reported desire to quit before and after the study and compare across groups.
Usability of the smartwatch and application | 12 weeks
  We will measure through self-report the usability participants experience while using the SmokeBeat application and smartwatch.
Usability of the smartwatch and application | 12 weeks
  We will measure through qualitative interviews the usability participants experience while using the SmokeBeat application and smartwatch.
Likability of the smartwatch and application | 12 weeks
  We will measure through self-report the likability participants experience while using the SmokeBeat application and smartwatch.
Likability of the smartwatch and application | 12 weeks
  We will measure through qualitative interviews the likability participants experience while using the SmokeBeat application and smartwatch.
Number of cigarettes smoked self-report | 12 weeks
  Number of cigarettes smoked in control vs. intervention group as measured by self-report.
Number of cigarettes smoked measured by smartwatch | 12 weeks
  Number of cigarettes smoked in control vs. intervention group as measured by the smartwatch.
Smoking cessation rate self-report | 12 weeks
  Quit rates in control vs. intervention group as measured by self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Buttenheim, PhD, MBA, Principal Investigator — University of Pennsylvania
Locations (1):
- Lancaster General Hospital, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Each participant will have a unique identifier to protect their confidentiality. Only pre-specified research coordinators will have access to identifiable participant information for contacting participants for follow-up.
  Only authorized personnel will have access to the data which will be maintained on encrypted hard-drives and destroyed after 7 years.

REFERENCES:
- [Background] McCallum DM, Fosson GH, Pisu M. Making the case for medicaid funding of smoking cessation treatment programs: an application to state-level health care savings. J Health Care Poor Underserved. 2014 Nov;25(4):1922-40. doi: 10.1353/hpu.2014.0171. PMID 25418250
- [Result] Centers for Disease Control and Prevention (CDC). The Health Consequences of Smoking: A Report of the Surgeon General. Atlanta: U.S. Department of Health and Human Services; 2004. U.S. Department of Health and Human Services. The Health Consequences of Smoking: A Report of the Surgeon General. Atlanta, GA: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention, National Center for Chronic Disease Prevention and Health Promotion, Office on Smoking and Health, 2004
- [Result] Salihu HM, Aliyu MH, Pierre-Louis BJ, Alexander GR. Levels of excess infant deaths attributable to maternal smoking during pregnancy in the United States. Matern Child Health J. 2003 Dec;7(4):219-27. doi: 10.1023/a:1027319517405. PMID 14682499
- [Result] Pregnancy Risk Assessment Monitoring System (PRAMS) and Smoking, Data from 2000-2011. http://www.cdc.gov/prams/pramstat/index.html
- [Result] Adams EK, Melvin CL, Raskind-Hood C, Joski PJ, Galactionova E. Infant delivery costs related to maternal smoking: an update. Nicotine Tob Res. 2011 Aug;13(8):627-37. doi: 10.1093/ntr/ntr042. Epub 2011 Jul 20. PMID 21778148
- [Result] Kornhauser M, Schneiderman R. How plans can improve outcomes and cut costs for preterm infant care. Manag Care. 2010 Jan;19(1):28-30. No abstract available. PMID 20131638
- [Result] Lumley J, Chamberlain C, Dowswell T, Oliver S, Oakley L, Watson L. Interventions for promoting smoking cessation during pregnancy. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD001055. doi: 10.1002/14651858.CD001055.pub3. PMID 19588322
- [Result] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Result] Prochaska JO, DiClemente CC. Stages and processes of self-change of smoking: toward an integrative model of change. J Consult Clin Psychol. 1983 Jun;51(3):390-5. doi: 10.1037//0022-006x.51.3.390. No abstract available. PMID 6863699
- [Result] Prochaska JO, DiClemente CC, Norcross JC. In search of how people change. Applications to addictive behaviors. Am Psychol. 1992 Sep;47(9):1102-14. doi: 10.1037//0003-066x.47.9.1102. PMID 1329589
- [Result] Weber EU, Johnson EJ, Milch KF, Chang H, Brodscholl JC, Goldstein DG. Asymmetric discounting in intertemporal choice: a query-theory account. Psychol Sci. 2007 Jun;18(6):516-23. doi: 10.1111/j.1467-9280.2007.01932.x. PMID 17576265
- [Derived] Joyce CM, Saulsgiver K, Mohanty S, Bachireddy C, Molfetta C, Steffy M, Yoder A, Buttenheim AM. Remote Patient Monitoring and Incentives to Support Smoking Cessation Among Pregnant and Postpartum Medicaid Members: Three Randomized Controlled Pilot Studies. JMIR Form Res. 2021 Sep 30;5(9):e27801. doi: 10.2196/27801. PMID 34591023